CLINICAL TRIAL: NCT04893772
Title: Observational Study to Assess Associations Between Daily Meal Timings, Appetite, Mood and Weight Loss in Individuals Completing a Commercial Intermittent Fasting Programme
Brief Title: Meal Timings, Appetite, Mood and Weight Loss in Individuals on a Commercial Intermittent Fasting Programme
Acronym: DASMA
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: LighterLife (UK) Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: DASMA_KCL
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2021-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Intermittent fasting — Three "fasting" days a week, whereby participants consume 600-800 kcal/day from 4 meal replacement products: breakfast, lunch, a snack and dinner. During the other 4 non-fasting "smart" days each week, participants are instructed to consume 2 x 300 kcal meals and 2 x 100 kcal snacks, from a selection of recipes, plus one meal of their own choosing.
  Other Names: LighterLife Fast

SUMMARY:
Although individuals following commercial intermittent fasting programmes consume meal replacement products during fasting days, further behavioural variables such as time of food consumption, sleep quality and duration, appetite and mood may significantly impact weight loss and intervention success. This project aims to assess behavioural patterns (dietary intake, sleep, meal timing, physical activity), mood and appetite on both fasting and non-fasting days and to investigate whether these are associated with weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Those responding to adverts on the LighterLife Fast Challenge social media channels will be asked if they would like to participate

Exclusion Criteria:

* Those without access to a smart phone or laptop will not be eligible to take part in the study due to the need to report variables daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults embarking on a commerical intermittent fasting weight loss programme
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight in kg | Change in body weight up to 12 weeks
  Weighed at home

SECONDARY OUTCOMES:
Sleep duration | Before weight loss programme (day 0)
  Pittsburg Sleep Quality Index (PSQI) questionnaire
Sleep quality | Before weight loss programme (day 0)
  Pittsburg Sleep Quality Index (PSQI) questionnaire
Physical activity | Before weight loss programme (day 0)
  Simple Physical Activity Questionnaire (SIMPAQ)
Meal timings | Before weight loss programme (day 0)
  Meal timings questionnaire
How hungry do you feel? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (I am not hungry at all) -100 (I have never been more hungry)
How satisfied do you feel? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (I am completely empty) -100 (I cannot eat another bite)
How full do you feel? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (not at all) -100 (totally full)
How much do you think you can eat? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (nothing at all) -100 (a lot)
Would you like to eat something sweet? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (yes very much) -100 (not at all)
Would you like to eat something salty? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (yes very much) -100 (not at all)
Would you like to eat something savoury? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (yes very much) -100 (not at all)
Would you like to eat something fatty? | Daily from day 1 up to 12 weeks
  Visual Analogue Scales, scale of 0 (yes very much) -100 (not at all)
Overall my mood is (very unpleasant to very pleasant) | Daily from day 1 up to 12 weeks
  Brief Mood Introspection Scale (BMIS), scale -10 to 10
Mindfulness - I was finding to difficult to stay focused on what I was doing | Weekly from week 1 up to 12 weeks
  Mindful Attention Awareness Scale (MASS), scale 0 (not at all) to 6 (very much)
Mindfulness - I was doing something without paying attention | Weekly from week 1 up to 12 weeks
  Mindful Attention Awareness Scale (MASS), scale 0 (not at all) to 6 (very much)
Mindfulness - I was preoccupied with the future or the past | Weekly from week 1 up to 12 weeks
  Mindful Attention Awareness Scale (MASS), scale 0 (not at all) to 6 (very much)
Mindfulness - I was doing something automatically without being aware of what I was doing | Weekly from week 1 up to 12 weeks
  Mindful Attention Awareness Scale (MASS), scale 0 (not at all) to 6 (very much)
Mindfulness - I was rushing through something without really being attentive to it. | Weekly from week 1 up to 12 weeks
  Mindful Attention Awareness Scale (MASS), scale 0 (not at all) to 6 (very much)
Height | Before weight loss programme (day 0)
  Height in cm
Dietary intake (macronutrients and energy) | Before weight loss programme (day 0)
  24 h recall x 2
Diet quality | Before weight loss programme (day 0)
  24 h recall x 2
Dietary intake (macronutrients and energy) | Non-fasting days: Weeks 1, 2, 3, 4, 8 and 12
  24 h recall x 4 (4 non-fasting days)
Diet quality | Non-fasting days: Weeks 1, 2, 3, 4, 8 and 12
  24 h recall x 4 (4 non-fasting days)
Meal replacement product choice | Fasting days: Weeks 1, 2, 3, 4, 8 and 12
  Question: Which meal replacement products did you consume?
Meal replacement product timings | Fasting days: Weeks 1, 2, 3, 4, 8 and 12
  Question: What time did you consume the meal replacement products?
Sleep duration | Daily from day 1 up to 12 weeks
  Question: How long did you sleep?
Sleep quality | Daily from day 1 up to 12 weeks
  Questions to rate quality of sleep
Physical activity | Daily from day 1 up to 12 weeks
  Question: Did you do any structured exercise today?
Alcohol use | Before weight loss programme (day 0)
  AUDIT questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutritional Sciences, King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No